CLINICAL TRIAL: NCT04593017
Title: Effect of Drops Containing Lactobacillus Reuteri (DSM 17938 and ATCC PTA 4659) on Plaque Acidogenicity and Other Caries Related Variables in Orthodontic Patients
Brief Title: On Probiotic, Dental Caries, and Orthodontic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 260-20
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Two groups matched in age and gender
Who Masked: Participant, Investigator
Masking Description: 3rd party will be involved in labeling the test and placebo samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Probiotic (Experimental): Probiotic contain active microorganism
  Interventions: Dietary Supplement: Active Probiotic
- Placebo Probiotic (Placebo Comparator): Probiotic with no active microorganism
  Interventions: Other: Placebo Probiotic

INTERVENTIONS:
Dietary Supplement: Active Probiotic — Lactobacillus Reuteri (DSM 17938 and ATCC PTA 4659
  Arms: Active Probiotic
Other: Placebo Probiotic — Placebo
  Arms: Placebo Probiotic

SUMMARY:
To investigate the short term effect of probiotic oil on plaque acidogenicity among orthodontic patients. Shortage on testing the effect of probiotic on Orthodontic patients can be seen on litterateurs making a gap of whether is product of help in preventing dental caries or not ?

DETAILED DESCRIPTION:
To investigate the short term effect of probiotic oil on plaque acidogenicity among orthodontic patients and to investigate the effect of probiotics on mutan streptococci and lactobacilli in plaque and saliva.

The null-hypothesis is that: The effect of probiotics would not differ from placebo-treated control group.

This product might decrease the chance of getting caries but also cooperation and cost effectiveness should be considered

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing bimaxillary fixed orthodontic treatment
* Number of S. mutans counts (>10.000 CFU/ml)
* Permanent dentition
* 3-12 months into the treatment (study from Sweden by Andrea)
* Medically healthy
* Not taking any medication
* Ability to understand the nature of the study and sign the consent form

Exclusion Criteria:

* Cleft lip and palate patients as well as handicapped and patients with mental impairments
* Systemic diseases or conditions that could interfere with our study (diabetes, immunosuppression diseases, pregnancy or ongoing therapy).
* History of probiotics/anti-inflammatory drugs taken during the last 4 weeks prior to baseline examination
* Local or general antimicrobial substances taken during the last 4 prior weeks prior to baseline examination
* Habitual consumers of xylitol chewing gums
* No active or untreated carious lesions and reported daily tooth brushing habit using fluoridated toothpaste

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Both Male and Female matched in age and gender
Enrollment: 28 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-21 (Estimated)

PRIMARY OUTCOMES:
Effect of Probiotic oil (drops) on plaque acidogenicity (pH) among orthodontic patients. | 3 weeks
  Changes in the plaque pH (acidic or alkaline) is an important factor among others in the cares process, in which an acidic environment will help the bacteria to accumulate along the tooth surface and starting the caries lesions.
  So, considering the plaque pH as a clinical variable to show the probiotic effect is considered to be of great value.

SECONDARY OUTCOMES:
Effect of Probiotics on Dental plaque | 3 weeks
  Plaque is an important aspect in caries detection, so the change in the plaque sample will show if the probiotic will help in the caries prevention during orthodontic treatment.
Effect of Probiotics on Saliva | 3 weeks
  The saliva composition which includes cariogenic bacteria (caries initiating bacteria) such as Streptococcus mutans and lactobacilli, is an important factor in caries detection, so saliva sample will show if the probiotic is helpful in caries prevention?

CONTACTS AND LOCATIONS:
Locations (1):
- Gothenburg university, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
This research planned for publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: As soon as we finish with the data collection and the manuscript writing, the data will be published online.

REFERENCES:
- [Derived] Alforaidi S, Bresin A, Almosa N, Lehrkinder A, Lingstrom P. Effect of drops containing Lactobacillus reuteri (DSM 17938 and ATCC PTA 5289) on plaque acidogenicity and other caries-related variables in orthodontic patients. BMC Microbiol. 2021 Oct 6;21(1):271. doi: 10.1186/s12866-021-02310-2. PMID 34615458